CLINICAL TRIAL: NCT00247520
Title: Two Center Evaluation of the Safety and Efficacy of Topical Nasal rEV131 Versus rEV131 Vehicle (Placebo)in the Prevention of the Signs and Symptoms of Allergic Rhinitis Induced by Nasal Allergen Challenge
Brief Title: Safety and Efficacy Study of rEV131 in Allergic Rhinitis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Evolutec Group (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EV-71-004
Record Dates: First submitted 2005-11-01; First posted 2005-11-02 (Estimated); Last update posted 2005-11-02 (Estimated); Status verified 2005-11

CONDITIONS: Hay Fever
Keywords: Seasonal allergic rhinitis (SAR), rhinoconjunctivitis, allergy
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Hypersensitivity

INTERVENTIONS:
Drug: topical nasal rEV131

SUMMARY:
The purpose of this study is to see whether rEV131 when given as a nasal spray in a single dose to each nostril is safe and can reduce the signs and symptoms of allergic rhinitis (hay fever) caused by an allergen challenge. All patients enrolled will be known to be allergic to ragweed pollen and will be given ragweed pollen extract in both nostrils 30 minutes after either rEV131 or innactive vehicle (placebo). The signs and symptoms (sneezing, itching, stuffiness and runny nose) will each be given a score from 0 to 3 by the patient and these will be added together and the combined scores from patients treated with rEV131 will be compared with those who received placebo.

DETAILED DESCRIPTION:
Hypothesis: rEV131, a histamine binding protein (derived from tick saliva) with an affinity for histamine 10 - 100 fold that of natural histamine receptors, might attenuate Nasal Allergen Challenge (NAC) induced allergic rhinitis.

Methods: Patients with known ragweed allergy will be screened to determine the minimal threshold concentration (PD30) of pollen extract that consistently induces the four key symptoms of allergic rhinitis: itch, sneezing, congestion and mucus production. A standardised system of TNSS scoring will be used. A total of 112 eligible patients will be randomised in double blind fashion to receive one of four concentrations of rEV131 (0.63, 1.25, 2.5 and 5.0 mg/ml) by nasal spray 30 minutes prior to NAC or placebo. Symptoms will be scored at 15, 30 and 45 minutes post NAC. Mean sum of symptom scores of all active medication treated patients will be compared with those of placebo treated patients. The primary analysis will be the sum of scores at 15 minutes post challenge for the optimum concentration of rEV131. Secondary outcome variables will include comparison of individual symptom and percentage of patients having a clinically significant response.

ELIGIBILITY:
Inclusion Criteria:

* a) Have a known past history of allergic rhinitis including allergy to ragweed pollen.

  b) Able and willing to give informed consent. c) Able and willing to follow all study related instructions. d) Able and willing to make all required visits. e) Aged between 18 and 80 years. f) Willing to avoid prohibited medications (see below). g) Has met at least one of the endpoints to allergen challenge at Visit 1
  1. Total symptom score of at least 6 OR
  2. ≥ 30% reduction in nasal volume in at least one side of the nose as measured by acoustic rhinometry AND total symptom score of at least 4.

     h) Has met endpoint to allergen challenge at Visit 2: Total symptom score of at least 4 from a possible total of 12.

     Exclusion Criteria:
* a) Patients with known exaggerated immuogenicity responses including severe asthma or peanut allergy.

  b) Patients with known allergy to ticks or severe reaction to arthropod venom (e.g. bee or wasp venom).

  c) Patients with known chronic sinusitis, deviated nasal septum or nasal polyposis.

  d) Patients having a total Baseline symptom score of >4 at Visit 1 (ie before the first nasal washout).

  e) Patients known or found to be allergic to pollens prevalent in the trial site locality during the period of the study (e.g. mountain cedar).

  f) Patients who have taken systemic or topical corticosteroids, long acting antihistamines or immunosuppressives within 4 weeks of selection (V1) or who take them within the course of the trial. Loratidine may not be taken within 10 days of entry. Short acting antihistamines may not be taken within 72 hours of entry except as comfort medication following nasal allergen challenge (oral antihistamines only). Patients excluded from the study for non-compliance with regard to prohibited medications but who have received one or more doses of the test medications will be included in the safety analysis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112
Dates: Start 2005-05; Study Completion 2005-08

PRIMARY OUTCOMES:
Sum of symptom scores at 15 minutes post allergen challenge

SECONDARY OUTCOMES:
Sum of symptom scores at 30 and 45 minutes post allergen challenge
Individual symptom scores at 15, 30 and 45 minutes post challenge
Pre and post treatment responder analysis
Change in nasal volume as assessed by acoustic rhinometry

CONTACTS AND LOCATIONS:
Overall Officials: Wynne H Weston-Davies, MB FRCS, Study Director — Evolutec Group plc
Locations (2):
- United States (2):
  - Diagnostics Research Group, San Antonio, Texas
  - Sylvana Research Associates, San Antonio, Texas